CLINICAL TRIAL: NCT04707664
Title: A Randomized Phase 2b Trial Evaluating Clinical Outcomes of Inhaled Sargramostim in High-risk Patients With Mild-moderate COVID-19
Brief Title: Sargramostim Use in COVID-19 to Recover Patient Health
Acronym: SCOPE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Partner Therapeutics, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PTX-001-003
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Results first posted 2023-02-06 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2022-12

CONDITIONS: Covid19; SARS-CoV Infection
Keywords: COVID-19; SARS-CoV2; sargramostim; Leukine; (recombinant human) GM-CSF; immune modulator; SCOPE
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Intervention Model Description: This Phase 2b, multicenter, placebo-controlled, double-blind study will randomize approximately 500 adult patients who are symptomatic with mild or moderate COVID-19 (as defined in the FDA Guidance Document: Covid-19: Developing Drugs and Biological Products for Treatment or Prevention, May 2020) who are at high risk for progression to more severe disease. Patients will be randomized in a 1:1 ratio to inhaled sargramostim plus standard of care (SOC) or placebo plus SOC. Enrollment of patients who have completed a COVID-19 vaccination regimen or participated in a COVID-19 vaccine clinical trial will be capped at approximately 100 patients.
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sargramostim Arm (Experimental): Day 1 - 5: Sargramostim treatment in addition to standard of care for COVID-19
  Interventions: Drug: Sargramostim
- Placebo Arm (Placebo Comparator): Day 1 - 5: Placebo treatment in addition to standard of care for COVID-19
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sargramostim — All patients randomized to the sargramostim treatment arm will be treated with 250 mcg inhaled sargramostim administered via a vibrating mesh nebulizer once daily for 5 days.
  Other Names: Leukine; GM-CSF
  Arms: Sargramostim Arm
Drug: Placebo — All patients in the control arm will receive an equivalent volume of inhaled placebo diluent administered via a vibrating mesh nebulizer once daily for 5 days.
  Arms: Placebo Arm

SUMMARY:
The purpose of this research is to understand if the study drug, also called sargramostim or Leukine®, can help prevent the worsening of COVID-19 when the study drug is inhaled. This study will also help researchers understand if inhaled sargramostim can help prevent visits to the emergency room or hospitalization, or death.

DETAILED DESCRIPTION:
This Phase 2b, multicenter, placebo-controlled, double-blind study will randomize approximately 500 adult patients who are symptomatic with mild or moderate COVID-19 (as defined in the FDA Guidance Document: Covid-19: Developing Drugs and Biological Products for Treatment or Prevention, May 2020) who are at high risk for progression to more severe disease. Patients will be randomized in a 1:1 ratio to inhaled sargramostim plus standard of care (SOC) or placebo plus SOC. Enrollment of patients who have completed a COVID-19 vaccination regimen or participated in a COVID-19 vaccine clinical trial will be capped at approximately 100 patients. All patients will be randomized to receive either 250 mcg of sargramostim or equivalent volume of placebo diluent. Treatment will be administered once daily for 5 days delivered via a vibrating mesh nebulizer. Patients will be followed for up to 60 days after start of treatment.

Sargramostim (Leukine) is a formulation of Granulocyte Macrophage Colony Stimulating Factor (GM-CSF), which is a critical cytokine for healthy pulmonary function. Detailed studies have shown that GM-CSF is necessary for alveolar macrophage (AM) maturation and maintenance. Although GM-CSF was discovered as a myelopoietic growth factor, it has diverse additional effects that both promote differentiation of myeloid precursors into neutrophils, monocytes, and dendritic cells and control function of mature myeloid cells. GM-CSF is also known to reverse immunoparalysis seen in sepsis, resulting in beneficial outcomes. In addition, GM-CSF prevents bacteremia in post influenza bacterial pneumonia through locally mediated improved lung antibacterial resistance and increased reactive oxygen species production by AMs. Pulmonary delivery of this GM-CSF has potential to reduce morbidity and mortality due to viral pneumonias, potentially including COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a positive laboratory diagnosis of SARS-CoV-2 infection by an antigen or a molecular test ≤5 days prior to randomization. The test should have been authorized by the relevant regulatory authority.
2. Have one or more of the following mild or moderate COVID-19 symptoms for ≤5 days prior to randomization:

   1. Fever or chills
   2. New onset or worsening cough
   3. Sore throat
   4. Malaise or fatigue
   5. Headache
   6. Muscle pain (myalgias) or body aches
   7. Gastrointestinal symptoms (e.g., nausea, vomiting, diarrhea)
   8. New onset or worsening shortness of breath or difficulty breathing
   9. Nasal congestion or runny nose
   10. New loss of taste (ageusia) and/or smell (anosmia). Note: any of these symptoms (ageusia, anosmia) alone or in combination cannot be used as the SOLE qualifying symptoms for enrollment.
3. At higher risk for progression to more severe COVID-19

   1. Age ≥ 60 years
   2. Age 18-59 years with a clinically stable medical history of at least 1 or more of the following conditions that could lead to severe COVID-19:

      * Chronic respiratory conditions such as asthma, chronic obstructive pulmonary disease (COPD), pulmonary fibrosis
      * Obesity with BMI ≥ 30 kg/m2
      * Cardiovascular disease
      * Sickle cell disease or thalassemia
      * Diabetes mellitus being managed with concomitant medications
      * Hypertension being managed with concomitant medications
      * Chronic kidney disease
4. Oxygen saturation by pulse oximeter > 93% on room air. Note: at altitudes of >4000 feet above sea level, oxygen saturation by pulse oximeter > 91% on room air is permitted
5. Negative pregnancy test (if woman of childbearing potential)
6. Females of childbearing potential and males with female partners of childbearing potential must agree to use acceptable contraceptive methods from screening to Day 28
7. The patient (or legally authorized decision maker) must give informed consent

Exclusion Criteria:

1. Hospitalized patients
2. Patients who have received or are receiving other treatments that are not approved/authorized by the relevant regulatory authority for the treatment of patients with mild or moderate COVID-19 in an outpatient setting
3. Patients enrolled in interventional clinical trials for other experimental therapies
4. Patients on chronic oxygen supplementation due to cardiopulmonary or other conditions
5. Patients with unstable comorbid conditions (e.g., decompensated congestive heart failure, COPD with exacerbation, current angina pectoris, uncontrolled diabetes mellitus, uncontrolled hypertension, uncontrolled asthma)
6. Patients with severe pulmonary comorbid conditions, including systemic steroid-dependent asthma, systemic steroid-dependent COPD, oxygen-dependent COPD, lung transplant, or cystic fibrosis
7. Patients who have received highly immunosuppressive therapy (to include systemic corticosteroids) or anti-cancer combination chemotherapy within 24 hours prior to first dose of study drug
8. Patients with known or suspected intolerance or hypersensitivity to sargramostim, or any component of the product
9. Patients who have previously experienced severe and unexplained side effects during aerosol delivery of any kind of medical product
10. Pregnant or breastfeeding females
11. Patients who, in the opinion of the Investigator, will not be able to comply with all the study procedures and visits as outlined in the schedule of events, including follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2022-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Garner, PhD, Study Director — Partner Therapeutics, Inc.
Locations (37):
- United States (34):
  - West Valley Research Clinic, LLC, Phoenix, Arizona
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Hope Clinical Research, Canoga Park, California
  - Benchmark Research, Colton, California
  - Synergy Healthcare, Bradenton, Florida
  - Invesclinic US, LLC., Fort Lauderdale, Florida
  - Indago Research & Health Center, Inc. (Subject Visits Only), Hialeah, Florida
  - Encore Medical Research, Hollywood, Florida
  - IMIC Inc., Palmetto Bay, Florida
  - Encore Medical Research of Weston, Weston, Florida
  - Gwinnett Research Institute, LLC, Buford, Georgia
  - Paramount Research Solutions, College Park, Georgia
  - TidalHealth Peninsula Regional, Inc., Salisbury, Maryland
  - Revive Research Institute, Inc., Farmington Hills, Michigan
  - Revival Research Institute, LLC., Sterling Heights, Michigan
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Great Plains Health, North Platte, Nebraska
  - Excel Clinical Research, Las Vegas, Nevada
  - Richmond University Medical Center, Staten Island, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Hometown Urgent Care and Research, Cincinnati, Ohio
  - Hometown Urgent Care and Research, Columbus, Ohio
  - Urgent Care Specialists, LLC DBA Hometown Urgent Care and Research, Dayton, Ohio
  - TruCare Internal Medicine and Infectious Disease, DuBois, Pennsylvania
  - Urgent Care Clinical Trials @ AFC Urgent Care - Easley, Easley, South Carolina
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - UCCT @ City Doc Urgent Care-McKinney, Dallas, Texas
  - Invesclinic US LLC, Edinburg, Texas
  - Dorrington Medical Associates, Houston, Texas
  - Encore Imaging & Medical Research, Houston, Texas
  - SMS Clinical Research, LLC, Mesquite, Texas
  - Novotrial Research Group, Pearland, Texas
  - Sun Research Institute, San Antonio, Texas
  - University of Utah Health, Salt Lake City, Utah
- Argentina (3):
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata, Buenos Aires
  - Instituto Medico de la Fundacion Estudios Clinicos, Rosario, Santa Fe Province
  - Sanatorio Santa Barbara, Buenos Aires

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sargramostim Arm | Placebo Arm
Started (All randomized patients) | 301 | 299
Full Analysis Set (Patients evaluated for efficacy) | 301 | 299
Safety Population (Patients who had at least 1 dose of assigned study treatment) | 297 | 290
Completed | 272 | 263
Not Completed | 29 | 36
Not completed — Adverse Event | 2 | 0
Not completed — Death | 1 | 2
Not completed — Withdrawal by Subject | 13 | 21
Not completed — Lost to Follow-up | 11 | 13
Not completed — Not treated | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sargramostim Arm | Placebo Arm | Total
Number analyzed (Participants) | 301 | 299 | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (15.38) | 43.5 (14.34) | 43.3 (14.86)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 136 | 138 | 274
  Female | 165 | 160 | 325
  Unknown | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 207 | 211 | 418
  Not Hispanic or Latino | 93 | 87 | 180
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 41 | 29 | 70
  White | 252 | 258 | 510
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 301 | 299 | 600
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI from 2 patients in the sargramostim arm and 2 patients in the placebo arm were not collected.
  kg/m^2
    number analyzed (Participants) | 299 | 297 | 596
    (all) | 32.3 (6.15) | 32.6 (6.03) | 32.5 (6.08)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Emergency Room Visit or Hospitalization, or Death by Day 28
Description: Percentage of patients who experience any emergency room visit or hospitalization, or death
Time Frame: 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sargramostim Arm | Placebo Arm
Number analyzed (Participants) | 301 | 299
Participants | 21 | 16

2. Secondary Outcome: Disease Progression Based on NIAID Score
Description: Proportion of patients with any progression of disease as determined by a ≥ 2-point increase from baseline in the National Institute of Allergy and Infectious Disease (NIAID) Ordinal Scale up to Day 28, and Day 60. The NIAID Ordinal Scale is a 1-8 scale and is an assessment of clinical status on a given study day. A score of 1 indicates the patient is not hospitalized and has no limitations on activities. A score of 8 indicates the patient has died.
Time Frame: Day 28 and Day 60
Population: The Full Analysis Set was used for analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Sargramostim Arm | Placebo Arm
Number analyzed (Participants) | 301 | 299
Participants
  By Day 28 | 14 | 14
  Day 29-60 | 0 | 0
  No COVID-19 progression | 287 | 285

3. Secondary Outcome: Time to Disease Progression Based on NIAID Score
Description: Time to progression of disease as determined by a ≥ 2-point increase in the NIAID ordinal scale up to Day 28, and Day 60. The NIAID ordinal scale is a 1-8 scale and is an assessment of clinical status on a given study day. A score of 1 indicates the patient is not hospitalized and has no limitations on activities. A score of 8 indicates the patient has died.
Time Frame: Day 28 and Day 60
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sargramostim Arm | Placebo Arm
Number analyzed (Participants) | 301 | 299
Days | NA [NA to NA] — The median time to progression of COVID-19 could not be calculated based on the small numbers of patients that progressed. | NA [NA to NA] — The median time to progression of COVID-19 could not be calculated based on the small numbers of patients that progressed.

4. Secondary Outcome: Change From Baseline in Overall Symptom Scores
Description: Change from baseline in overall symptom score as measured by the Symptom Score Questionnaire on Day 7, Day 14 and Day 28. The overall symptom score is the sum of 14 individual symptom scores from Symptom Score Questionnaire. Individual symptom scores correspond to the following responses: None = 0, Mild = 1, Moderate = 2, Severe = 3; None = 0, 1-2 times = 1, 3-4 times = 2, 5 or more times = 3; Same as usual = 0, Less than usual = 1, No sense = 2. The lowest score could be 0, and the highest score could be 42. Patients with higher scores have more severe symptoms from COVID-19.
Time Frame: Day 7, 14, and 28
Population: The Full Analysis Set was used
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sargramostim Arm | Placebo Arm
Number analyzed (Participants) | 301 | 299
score on a scale
  Day 7 | -7.7 (7.02) | -6.7 (7.33)
  Day 14 | -11.7 (6.62) | -10.6 (7.35)
  Day 28 | -13.8 (6.69) | -13.3 (7.19)

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events up to Day 60
Time Frame: 60 days
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Sargramostim Arm | Placebo Arm
Number analyzed (Participants) | 297 | 290
Participants | 59 | 67

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 60 days
Description: Evaluation of safety and all-cause mortality was conducted with the Safety Population, having at least 1 dose of study treatment. Worsening of COVID-19 signs and symptoms were exempt from AE reporting, unless related to study treatment administration or judged to be more severe than expected.
Arm/Group | Sargramostim Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 1/297 | 2/290
Serious Adverse Events (participants affected / at risk) | 13/297 | 11/290
Other Adverse Events (participants affected / at risk) | 46/297 | 56/290
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Sargramostim Arm (N=297) | Placebo Arm (N=290)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 4 (4) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 2 (2)
Appendicitis (Infections and infestations) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
SARS-CoV-2 sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Exposure during pregnancy (Injury, poisoning and procedural complications) | 1/164 (1) | 0/154 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Sargramostim Arm (N=297) | Placebo Arm (N=290)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Swollen lymph nodes
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) — Dizziness
Vision blurred (Eye disorders) | 1 (1) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 1 (1) — Eye redness
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) — increased tear production
Ocular hyperaemia (Eye disorders) | 1 (1) | 0 (0) — Eye redness
Vomiting (Gastrointestinal disorders) | 3 (4) | 4 (4)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 0 (0) — Tongue pain
Tongue discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 2 (2) | 1 (1)
Fatigue (General disorders) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (3) — Fever
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) — swelling in extremities
Hepatosplenomegaly (Hepatobiliary disorders) | 1 (1) | 0 (0) — Enlarged liver and spleen
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2)
Otitis media acute (Infections and infestations) | 1 (1) | 1 (1) — ear infection
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0) — sore throat
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) — Stye
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 1/164 (1) | 0/154 (0) — Yeast infection
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 2 (2) | 2 (2)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Fibrin D dimer increased (Investigations) | 2 (2) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 1 (1)
Neutrophil count increased (Investigations) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood lactate dehydrogenase abnormal (Investigations) | 0 (0) | 1 (1)
Blood potassium increased (Investigations) | 0 (0) | 1 (1)
Serum ferritin increased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (6)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Haemochromatosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 6 (6)
Paraesthesia (Nervous system disorders) | 2 (2) | 4 (4)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Acute sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-08-23): https://cdn.clinicaltrials.gov/large-docs/64/NCT04707664/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-13): https://cdn.clinicaltrials.gov/large-docs/64/NCT04707664/SAP_001.pdf